CLINICAL TRIAL: NCT03596450
Title: Long Term Comparative Effectiveness of Once Weekly Semaglutide Versus Standard of Care in a Real World Adult US Population With Type 2 Diabetes - a Randomized Pragmatic Clinical Trial
Brief Title: Long Term Comparative Effectiveness of Once Weekly Semaglutide Versus Standard of Care in a Real World Adult US Population With Type 2 Diabetes - a Randomized Pragmatic Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4416; U1111-1207-6474 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide subcutaneously (s.c.) in addition to metformin monotherapy as treatment intensification in the course of routine clinical practice. Participants will be followed for 2 years, regardless of changes in antidiabetic treatment over the course of the study.
  Interventions: Drug: Semaglutide
- Standard of care (Active Comparator): Participants will receive standard of care in addition to metformin monotherapy as treatment intensification in the course of routine clinical practice. Participants will be followed for 2 years, regardless of changes in antidiabetic treatment over the course of the study.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Semaglutide — Participants will be prescribed commercially available semaglutide s.c. and will be instructed to initiate treatment with semaglutide s.c. according to the approved label. The study doctor will determine the intended maintenance dose of semaglutide, as well as changes to the maintenance dose thereafter.
  Arms: Semaglutide
Drug: Standard of care — Participants will receive standard of care, defined as commercially available oral or injectable antidiabetic medication other than semaglutide. Participants will be prescribed and instructed to initiate commercially available antidiabetic medication according to the approved label and, if relevant for the specific antidiabetic medication, adjusted at the discretion of the study doctor.
  Arms: Standard of care

SUMMARY:
The main purpose of this study is to compare the effects of semaglutide (Ozempic®) with the effects of other treatments for type 2 diabetes in a normal practice setting. The participant will be assigned by chance (like flipping a coin) to one of the following treatment groups: Group 1: semaglutide (Ozempic®) (by injection into skin) Group 2: standard of care antidiabetic medication (oral or injectable). The participant has an equal chance of being in either of the treatment groups. Neither the participant nor the study doctor or study staff will be able to pick which group the participant is in, but the participant will know which study drug the participant has been assigned to. The study doctor will provide the participant with a prescription for the study diabetes medication based on the treatment group the participant is assigned. The participation will last about 2 years.

ELIGIBILITY:
Inclusion Criteria:-

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study.
* Male or female, age 18 years or older at the time of signing informed consent.
* Type 2 diabetes mellitus diagnosis.
* Treatment with either 1 or 2 oral antidiabetic medications.
* Current member of a commercial or Medicare health plan with pharmacy benefits.
* Recorded HbAlc value within the last 90 days prior to randomization.
* Further intensification with an additional antidiabetic oral or injectable medication is indicated to achieve glycemic target at the discretion of the study physician according to approved labelling.

Exclusion Criteria:

* Previous randomization in this study
* Treatment with more than 2 oral antidiabetic medications, oral semaglutide, or any injectable medication in a period of 30 days before the day of eligibility assessment. Temporary/emergency use of any type of insulin is allowed, as is prior insulin treatment for gestational diabetes.
* Contraindications to semaglutide according to the Food and Drug Administration approved label.
* Female who is pregnant, breastfeeding or intends to become pregnant
* Participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1278 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (122):
- United States (121):
  - American Clinical Trials, Buena Park, California
  - St. Jos Heritage Hlthcr_Fllrtn, Fullerton, California
  - SC Clinical Research, Inc., Garden Grove, California
  - New Hope Consulting & Clinical Trials, Lancaster, California
  - OM Research LLC, Lancaster, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Pacific Medical Center, Milpitas, California
  - Facey Medical Foundation, Mission Hills, California
  - Monterey Endocrine & Diabetes Institute, Inc, Monterey, California
  - Do-Eun Lee, Napa, California
  - Format Medical Research, Oxnard, California
  - Joselito C Cabaccan, MD, San Jose, California
  - Premier Medical Center, Inc., Toluca Lake, California
  - Adnab Research/Prestige Care Physician, Torrance, California
  - Altura Centers For Health, Tulare, California
  - Tariq Javed, MD Inc., Visalia, California
  - Endocrinology & Diabetes Specialists, Walnut Creek, California
  - University of Colorado Hospital, Denver, Colorado
  - Denver Endocrinology Diabetes and Thyroid Center, Englewood, Colorado
  - ProHealth Physicians/OptumCare, Bristol, Connecticut
  - Western Connecticut Health Network_Danbury, Danbury, Connecticut
  - Endocrine Associates of Connecticut, Hamden, Connecticut
  - Ismail Tarkhan MD, Milford, Connecticut
  - Steven L. Saunders MD LLC, Milford, Connecticut
  - The Kaufmann Clinic, Inc., Atlanta, Georgia
  - Primary Care Research, Atlanta, Georgia
  - Southern Family Medical Center, Augusta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Gwinnett Research Insti/Buford Family Pract Urgent Care Ctr, Buford, Georgia
  - Centricity Research, Columbus, Georgia
  - Medical Care of LaGrange, La Grange, Georgia
  - Beaver Ruin Primary Care, Lilburn, Georgia
  - Privia Medical Group of Georgia LLC, Locust Grove, Georgia
  - DC Research Works, Marietta, Georgia
  - Urban Family Practice Assoc, Marietta, Georgia
  - Atlanta Center for Clinical Research, Roswell, Georgia
  - Sandersville Family Practice, Sandersville, Georgia
  - Meridian Clin Res, LLC, Savannah, Georgia
  - Family Health Care Center, Statesboro, Georgia
  - Eagles Landing Diabetes/Endocrinology, Stockbridge, Georgia
  - Herman Clinical Research LLC, Suwanee, Georgia
  - Sugarloaf Medical, PC, Suwanee, Georgia
  - East Georgia Healthcare Center Inc, Swainsboro, Georgia
  - Coastal Care Medical Clinic, Waycross, Georgia
  - St. Vincent Research Institute, Anderson, Indiana
  - American Health Network of Indiana, LLC_Avon_0, Avon, Indiana
  - Adams County Family Physicians, Berne, Indiana
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Associated Surgeons & Physicians LLC, Fort Wayne, Indiana
  - American Health Network of IN LLC_Franklin, Franklin, Indiana
  - American Health Network of Indiana, LLC_Greenfield, Greenfield, Indiana
  - La Porte County Institute For Clinical Research, Michigan City, Indiana
  - Beacon Medical Group Swartz-Weikamp, Mishawaka, Indiana
  - American Health Network of IN LLC, Muncie, Indiana
  - American Health Network of Indiana, LLC, New Albany, Indiana
  - Reid Endocrinology Center, Richmond, Indiana
  - Regional Endorine and Diabetes Associates, Ashland, Kentucky
  - Tri State Primary Caregrayson Health Park, Ashland, Kentucky
  - St Elizabeth Physicians Heart, Covington, Kentucky
  - The Endocrine & Diabetes Center, Owensboro, Kentucky
  - Paris Family Physicians PLLC, Paris, Kentucky
  - Gaurang B. Shah, MD, Richmond, Kentucky
  - WCMP Family Medicine, Belfast, Maine
  - Tri-County Research, Inc., Sterling Heights, Michigan
  - Diabetes & Endo Specialists Inc, Chesterfield, Missouri
  - University Of Missouri - Columbia, Columbia, Missouri
  - Jefferson City Medical Group, PC, Jefferson City, Missouri
  - Trinity Healthcare, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - South County Endocrinology and Obesity Medicine, LLC, St Louis, Missouri
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Albany Medical College - Endo, Albany, New York
  - Prominis Medical Services PC, Brooklyn, New York
  - Northwell Health Div of Endo, Great Neck, New York
  - Advanced Internal Medicine Group, Great Neck, New York
  - NYC Research, Inc., New York, New York
  - NYU Grossman School of Med, New York, New York
  - EDOC LLP, Yonkers, New York
  - OnSite Clinical Solutions, LLC_Charlotte_0, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC_Charlotte, Charlotte, North Carolina
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - Catherine LaRuffa, M.D., Inc., Blanchester, Ohio
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Medical Frontiers, LLC, Carlisle, Ohio
  - University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio
  - Central Ohio Clinical Research LLC, Columbus, Ohio
  - Centricity Research, Columbus, Ohio
  - Franklin Family Practice, Franklin, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Functional Endocrinology, Mason, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Primary Care Research South, Inc, McMurray, Pennsylvania
  - Preferred Primary Care Physicians_Pittsburgh, Pittsburgh, Pennsylvania
  - Athens Medical Group, Athens, Tennessee
  - PMG Research of Bristol, Bristol, Tennessee
  - Murphy Research Center, Humboldt, Tennessee
  - Ascend Research Centers, Inc., McMinnville, Tennessee
  - Christus Trinity Clinic Hill Country Landa, New Braunfels, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - The Endocrinology Group, Arlington, Virginia
  - Chatham Family Medical Center, Chatham, Virginia
  - Swift Creek Family Care, Colonial Heights, Virginia
  - Lawson Family Medicine & Aesthetics, Daleville, Virginia
  - Privia Medical Group LLC, Danville, Virginia
  - Seven Corners Medical, Falls Church, Virginia
  - Hampton Family Practice, Hampton, Virginia
  - Medical Associates of Central Virginia, Inc., Lynchburg, Virginia
  - C. Lee Ginsburgh, Newport News, Virginia
  - Family Medicine Healthcare, Portsmouth, Virginia
  - Family Health Clinic, Radford, Virginia
  - Halifax Internal Medicine, South Boston, Virginia
  - Hampton Roads Center for Clinical Research, Suffolk, Virginia
  - Endocrinology Consultants, Virginia Beach, Virginia
  - Corporation Lane Research Center, Virginia Beach, Virginia
  - Piedmont Family Practice PLC, Warrenton, Virginia
  - Family Care of Williamsburg, Williamsburg, Virginia
  - St. Vincent Hosp-Prevea Health, Green Bay, Wisconsin
  - Ascension Medical Group- Germantown Clinic, Milwaukee, Wisconsin
  - Medical College of Wisconsin & Zablocki VAMC, Milwaukee, Wisconsin
- Western University Medical Center at WU of Health Sciences, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Buse JB, Nordahl Christensen H, Harty BJ, Cziraky MJ, Willey VJ, Skibsted S. Long-term comparative effectiveness of once-weekly semaglutide versus alternative treatments in a real-world US adult population with type 2 diabetes: a randomized pragmatic clinical trial. BMJ Open Diabetes Res Care. 2025 Oct 15;13(5):e005161. doi: 10.1136/bmjdrc-2025-005161. PMID 41093600
- [Derived] Buse JB, Nordahl Christensen H, Harty BJ, Mitchell J, Soule BP, Zacherle E, Cziraky M, Willey VJ. Study design and baseline profile for adults with type 2 diabetes in the once-weekly subcutaneous SEmaglutide randomized PRAgmatic (SEPRA) trial. BMJ Open Diabetes Res Care. 2023 May;11(3):e003206. doi: 10.1136/bmjdrc-2022-003206. PMID 37137527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 138 sites in the United States.
Pre-assignment Details: A total of 1,278 participants were randomized 1:1 to receive either semaglutide or standard of care (SOC).
Groups:
- Semaglutide: Participants received semaglutide subcutaneous (s.c.) injection once weekly in addition to up to 2 oral antidiabetic medications as treatment intensification for 2 years. Medication dose and dose escalation was at the discretion of the study physician according to routine practice for medications for glycemic control in participants.
- Standard of Care: Participants received standard of care (any commercially available oral or injectable antidiabetic medication, excluding semaglutide) in addition to up to 2 oral antidiabetic medications as treatment intensification for 2 years. Medication dose and dose escalation was at the discretion of the study physician according to routine practice for medications for glycemic control in participants.
Period: Overall Study
Arm/Group | Semaglutide | Standard of Care
Started | 644 | 634
Completed | 463 | 447
Not Completed | 181 | 187
Not completed — Death | 9 | 9
Not completed — Protocol Violation | 18 | 26
Not completed — Lost to Follow-up | 50 | 56
Not completed — Adverse Event | 14 | 7
Not completed — Withdrawal by Subject | 38 | 36
Not completed — Accidentally Randomized | 2 | 0
Not completed — Other reasons | 48 | 53
Not completed — Pregnancy | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants analyzed according to the treatment group to which they were assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Standard of Care | Total
Number analyzed (Participants) | 644 | 634 | 1278
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.47 (11.305) | 57.24 (10.982) | 57.36 (11.142)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data for one participant is missing in the Semaglutide arm.
  Participants
    number analyzed (Participants) | 643 | 634 | 1277
    Female | 309 | 276 | 585
    Male | 334 | 358 | 692
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 57 | 114
  Not Hispanic or Latino | 586 | 577 | 1163
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 517 | 487 | 1004
  Black or African American | 90 | 99 | 189
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  American Indian or Alaska Native, Asian | 16 | 27 | 43
  Other | 17 | 19 | 36
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Glycosylated Haemoglobin (HbA1c) Less Than 7.0 Percentage (%) (53 Millimoles Per Mole [mmol/Mol]) at Year 1 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0 % (53 mmol/mol) at year 1 is presented. Yes: number of participants who achieved HbA1c less than 7.0 % at year 1; No: number of participants who did not achieve HbA1c less than 7.0 % at year 1.
Time Frame: At year 1
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 430 | 462
Participants
  Yes | 244 | 226
  No | 186 | 236
Statistical Analysis 1: Comparison: Semaglutide vs Standard of Care; Estimate and p-value are based on logistic regression model with logit link function, treatment as categorical effect, and baseline HbA1c as covariate; Test type: Superiority; p = 0.033, Regression, Logistic; Treatment effect = 1.36, 95% CI 2-sided [1.03 to 1.79]

2. Secondary Outcome: Change in HbA1c (Percentage-point [%-Point]) From Baseline to Year 1
Description: Change in HbA1c from baseline to year 1 is presented in %-point.
Time Frame: Baseline (less than or equal to 90 days prior to randomization at week 0), year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage-point of HbA1c
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 430 | 461
Percentage-point of HbA1c | -1.46 (1.669) | -1.14 (1.707)

3. Secondary Outcome: Number of Participants With Glycosylated Haemoglobin (HbA1c) Less Than 7.0% (53 Millimoles Per Mole [mmol/Mol]) at Year 2 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0 % (53 mmol/mol) at year 2 is presented. Yes: number of participants who achieved HbA1c less than 7.0 % at year 2; No: number of participants who did not achieve HbA1c less than 7.0 % at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 374 | 374
Participants
  Yes | 209 | 162
  No | 165 | 212

4. Secondary Outcome: Change in HbA1c (Percentage-point [%-Point]) From Baseline to Year 2
Description: Change in HbA1c from baseline to year 2 is presented in percentage-point.
Time Frame: Baseline (less than or equal to 90 days prior to randomization at week 0), year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage-point of HbA1c
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 374 | 373
Percentage-point of HbA1c | -1.45 (1.723) | -0.98 (1.767)

5. Secondary Outcome: Number of Participants Who Attained Individualized HbA1c Target at Year 1 (Yes/No)
Description: Number of participants who attained individualized HbA1c target at year 1 is presented. Study physicians set and documented an individualized HbA1c target for participants prior to randomization based on their clinical judgement and knowledge of the participant. Yes: number of participants who achieved individualized HbA1c target attained at year 1; No: number of participants who did not achieve individualized HbA1c target attained at year 1
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 430 | 462
Participants
  Yes | 216 | 170
  No | 214 | 292

6. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) or At Least 1% Point Improvement in HbA1c Compared to Baseline at Year 1 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) or at least 1% point improvement in HbA1c compared to baseline at year 1 is presented. Yes: number of participants who achieved HbA1c less than 7.0% or at least 1% point improvement in HbA1c compared to baseline at year 1; No: number of participants who did not achieve HbA1c less than 7.0% or at least 1% point improvement in HbA1c compared to baseline at year 1
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 430 | 462
Participants
  Yes | 321 | 301
  No | 109 | 160
  Data missing | 0 | 1

7. Secondary Outcome: Number of Participants With HbA1c Target Attainment Per Healthcare Effectiveness Data and Information Set (HEDIS) Criteria at Year 1 (Yes/No)
Description: Number of participants who achieved HbA1c target attainment per HEDIS criteria (less than 8.0% if age ≥ 65 years or with defined comorbidities, otherwise less than 7.0%) at year 1 is presented. Yes: Number of participants who achieved HbA1c target attainment per HEDIS criteria at year 1; No: Number of participants who did not achieve HbA1c target attainment per HEDIS criteria at year 1
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 95 | 98
Participants
  Yes | 64 | 53
  No | 31 | 45

8. Secondary Outcome: Change in Body Weight (in Pounds) From Baseline to Year 1
Description: Change in body weight (in pounds) from baseline to year 1 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 458 | 461
Pounds (lbs) | -9.8 (21.15) | -5.4 (20.70)

9. Secondary Outcome: Percentage Change in Body Weight From Baseline to Year 1
Description: Percentage change in body weight from baseline to year 1 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 458 | 461
Percentage change in body weight | -3.93 (11.092) | -2.02 (8.924)

10. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Year 1
Description: Change in SBP from baseline to year 1 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 456 | 457
Millimeters of mercury (mmHg) | -2.3 (16.40) | -1.8 (16.34)

11. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline to Year 1
Description: Change in DBP from baseline to year 1 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 456 | 457
mmHg | -1.6 (10.08) | -0.9 (9.79)

12. Secondary Outcome: Time to First Study Drug Discontinuation During 2 Years
Description: Time to first study drug discontinuation during 2 years is presented. First study drug discontinuation=date of the first time a patient is not taking study drug as defined.
Time Frame: Week 0 to year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 634 | 621
Years | 1.36 (0.853) | 1.54 (0.719)

13. Secondary Outcome: Time to First Treatment Intensification (Add-on) or Change (Switch) After Randomization During 2 Years
Description: Time to first treatment intensification (add-on) or change (switch) after randomization during 2 years is presented.
Time Frame: Week 0 to year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 575 | 550
Years | 1.55 (0.731) | 1.43 (0.742)

14. Secondary Outcome: Percentage of Medication Possession Ratio (MPR) for Study Drug Medication Adherence for the First Year of the Study
Description: Percentage of MPR for study drug medication adherence for the first year of the study is presented. Medication adherence referred to a participant's conformance to the provider's recommendation with respect to timing, dosage, and frequency of medication taken during the prescribed length of time. The MPR was used to assess adherence. MPR was calculated as follows: MPR (%) = Sum of days supply for all prescription fills*100/Total number of days in time period. MPR was capped at 100%. MPR was calculated from pharmacy claims data and irrespective of adherence to randomized treatment or changes to antidiabetic treatment.
Time Frame: Week 0 to year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of MPR
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 135 | 134
Percentage of MPR | 53.1 (40.9) | 55.8 (41.2)

15. Secondary Outcome: Number of Hypoglycemic Episodes Leading to an Inpatient Admission or Emergency Room (ER) Encounter From Baseline to Year 2
Description: Number of hypoglycemic episodes leading to an inpatient admission or emergency room (ER) encounter from baseline to year 2 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 644 | 634
Episodes | 2 | 1

16. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire, Change Version (DTSQc), Total Treatment Satisfaction Score Measured at Year 1
Description: DTSQc total treatment satisfaction score measured at year 1 is presented. The DTSQc provides a measure of how satisfied participants are with their current diabetes treatment compared with previous treatment. It consists of 8 questions, which are to be answered on a Likert scale from -3 to +3 (-3 = much less satisfied now to +3 = much more satisfied now), with 0 (midpoint), representing no change. Six questions are summed to produce a total treatment satisfaction score. The remaining two questions concern perceived frequency of hyperglycemia and perceived frequency of hypoglycemia, respectively. The DTSQc total treatment satisfaction score ranges from -18 to +18, with higher scores associated with greater treatment satisfaction.
Time Frame: At year 1
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for this outcome measure. Analysis is based only on participants with available data for DTSQ at the dedicated study visit including measurements irrespective of whether participants discontinued study drug or not.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 447 | 460
Scores on a scale | 13.5 (5.28) | 12.8 (5.82)

17. Secondary Outcome: DTSQc, Total Treatment Satisfaction Score Measured at Year 2
Description: DTSQc total treatment satisfaction score measured at year 2 is presented. The DTSQc provides a measure of how satisfied participants are with their current diabetes treatment compared with previous treatment. It consists of 8 questions, which are to be answered on a Likert scale from -3 to +3 (-3 = much less satisfied now to +3 = much more satisfied now), with 0 (midpoint), representing no change. Six questions are summed to produce a total treatment satisfaction score. The remaining two questions concern perceived frequency of hyperglycemia and perceived frequency of hypoglycemia, respectively. The DTSQc total treatment satisfaction score ranges from -18 to +18, with higher scores associated with greater treatment satisfaction.
Time Frame: At year 2
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 388 | 380
Scores on a scale | 13.2 (6.24) | 12.2 (5.87)

18. Secondary Outcome: Change From Baseline in Short Form 12-Item Version 2 Survey (SF-12 v2), Physical Component Summary (PCS-12) Score at Year 1
Description: Change from baseline in SF-12 v2, PCS-12 score at year 1 is presented. The SF-12 v2 is a 12-item generic health-related quality of life measure that assesses physical and mental functioning. The items were scored using the scoring software. It contains two summary scores: Physical Component Summary (PCS) Score and Mental Component Summary (MCS) Score. The scores are norm-scored such that the scores range from 0-100 with a mean of 50 and standard deviation of 10. A higher score is associated with better quality of life and a lower score, poorer quality of life.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for this outcome measure. Analysis is based only on participants with available data for SF-12 at dedicated study visit including measurements irrespective of whether participants discontinued study drug or not.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 439 | 449
Scores on a scale | 2.8 (8.20) | 2.3 (7.60)

19. Secondary Outcome: Change From Baseline in SF-12 v2, PCS-12 Score at Year 2
Description: Change from baseline in SF-12 v2, PCS-12 score at year 2 is presented. The SF-12 v2 is a 12-item generic health-related quality of life measure that assesses physical and mental functioning. The items were scored using the scoring software. It contains two summary scores: Physical Component Summary (PCS) Score and Mental Component Summary (MCS) Score. The scores are norm-scored such that the scores range from 0-100 with a mean of 50 and standard deviation of 10. A higher score is associated with better quality of life and a lower score, poorer quality of life.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 383 | 376
Scores on a scale | 2.6 (8.68) | 2.4 (7.99)

20. Secondary Outcome: Change From Baseline in SF-12 v2, Mental Component Summary (MCS-12) Score at Year 1
Description: Change from baseline in SF-12 v2, MCS-12 score at year 1 is presented. The SF-12 v2 is a 12-item generic health-related quality of life measure that assesses physical and mental functioning. The items were scored using the scoring software. It contains two summary scores: PCS Score and MCS Score. The scores are norm-scored such that the scores range from 0-100 with a mean of 50 and standard deviation of 10. A higher score is associated with better quality of life and a lower score, poorer quality of life.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 439 | 449
Scores on a scale | 2.4 (8.54) | 1.1 (8.17)

21. Secondary Outcome: Change From Baseline in SF-12 v2, MCS-12 Score at Year 2
Description: Change from baseline in SF-12 v2, MCS-12 score at year 2 is presented. The SF-12 v2 is a 12-item generic health-related quality of life measure that assesses physical and mental functioning. The items were scored using the scoring software. It contains two summary scores: PCS Score and MCS Score. The scores are norm-scored such that the scores range from 0-100 with a mean of 50 and standard deviation of 10. A higher score is associated with better quality of life and a lower score, poorer quality of life.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 383 | 376
Scores on a scale | 2.4 (8.43) | 0.2 (9.31)

22. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment, General Health Questionnaire (WPAI-GH) Absenteeism (Work Time Missed) Score at Year 1
Description: Change from baseline in WPAI-GH Absenteeism (work time missed) score at year 1 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work/reduced on-the-job effectiveness), Work productivity loss (overall work impairment/absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for this outcome measure. Analysis is based only on participants with available data for WPAI-GH at the dedicated study visit including measurements irrespective of whether participants discontinued study drug or not.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 236 | 241
Scores on a scale | -1.5 (21.39) | 0.9 (14.39)

23. Secondary Outcome: Change From Baseline in WPAI-GH Absenteeism (Work Time Missed) Score at Year 2
Description: Change from baseline in WPAI-GH Absenteeism (work time missed) score at year 2 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work/reduced on-the-job effectiveness), Work productivity loss (overall work impairment/absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 204 | 200
Scores on a scale | -2.1 (22.86) | 0.0 (14.15)

24. Secondary Outcome: Change From Baseline in WPAI-GH Presenteeism (Impairment at Work/Reduced On-the-job Effectiveness) Score at Year 1
Description: Change from baseline in WPAI-GH Presenteeism (Impairment at Work/Reduced On-the-job Effectiveness) score at year 1 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work / reduced on-the-job effectiveness), Work productivity loss (overall work impairment / absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 230 | 238
Scores on a scale | -5.1 (24.31) | -4.5 (22.25)

25. Secondary Outcome: Change From Baseline in WPAI-GH Presenteeism (Impairment at Work/Reduced On-the-job Effectiveness) Score at Year 2
Description: Change from baseline in WPAI-GH Presenteeism (Impairment at Work/Reduced On-the-job Effectiveness) score at year 2 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work / reduced on-the-job effectiveness), Work productivity loss (overall work impairment / absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 196 | 198
Scores on a scale | -6.0 (24.30) | -3.8 (24.89)

26. Secondary Outcome: Change From Baseline in WPAI-GH Work Productivity Loss (Overall Work Impairment/Absenteeism Plus Presenteeism) Score at Year 1
Description: Change from baseline in WPAI-GH work productivity loss (overall work impairment/absenteeism plus presenteeism) score at year 1 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work / reduced on-the-job effectiveness), Work productivity loss (overall work impairment / absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 229 | 238
Scores on a scale | -4.8 (25.64) | -4.5 (24.79)

27. Secondary Outcome: Change From Baseline in WPAI-GH Work Productivity Loss (Overall Work Impairment/Absenteeism Plus Presenteeism) Score at Year 2
Description: Change from baseline in WPAI-GH work productivity loss (overall work impairment/absenteeism plus presenteeism) score at year 2 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work / reduced on-the-job effectiveness), Work productivity loss (overall work impairment / absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 196 | 198
Scores on a scale | -6.4 (25.18) | -4.0 (25.89)

28. Secondary Outcome: Change From Baseline in WPAI-GH Activity Impairment Score at Year 1
Description: Change from baseline in WPAI-GH activity impairment score at year 1 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work/reduced on-the-job effectiveness), Work productivity loss (overall work impairment/absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 435 | 445
Scores on a scale | -6.7 (27.91) | -3.7 (27.15)

29. Secondary Outcome: Change From Baseline in WPAI-GH Activity Impairment Score at Year 2
Description: Change from baseline in WPAI-GH activity impairment score at year 2 is presented. The WPAI-GH yields four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work/reduced on-the-job effectiveness), Work productivity loss (overall work impairment/absenteeism plus presenteeism), and Activity Impairment. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes (percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health, percent activity impairment due to health).
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 379 | 375
Scores on a scale | -5.8 (27.51) | -3.1 (28.03)

30. Secondary Outcome: All Cause Healthcare Resource Utilization (HCRU): Mean Number of Inpatient Admissions Per Participant From Baseline to Year 2
Description: All cause healthcare resource utilization - mean number of inpatient admissions per participant from baseline to year 2 is presented.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for this outcome measure. Analysis is based only on participants with available data for HCRU at dedicated study visit including measurements irrespective of whether participants discontinued study drug or not.
Measure: Mean (Standard Deviation); unit: inpatient admissions
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
inpatient admissions | 0.20 (0.55) | 0.25 (0.90)

31. Secondary Outcome: All Cause HCRU: Mean Cumulative Length of Stay for Inpatient Admissions Per Participant From Baseline to Year 2
Description: All cause HCRU - mean cumulative length of stay for inpatient admissions per participant from baseline to year 2 is presented. Cumulative inpatient length of stay is the sum of the length of stay of all inpatient admissions a participant experiences from baseline to year 2.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for this outcome measure. Analysis is based only on participants with available data for HCRU at dedicated study visit including measurements irrespective of whether participants discontinued study drug or not. It is only calculated for participants with at least one inpatient admission.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 16 | 16
Days | 4.7 (3.4) | 7.7 (12.1)

32. Secondary Outcome: All Cause HCRU: Mean Number of Emergency Room (ER) Encounters Per Participant From Baseline to Year 2
Description: All cause HCRU - mean number of emergency room (ER) encounters per participant from baseline to year 2 is presented.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: ER encounters
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
ER encounters | 0.72 (2.01) | 0.29 (0.77)

33. Secondary Outcome: All Cause HCRU: Mean Number of Outpatient Encounters Per Participant From Baseline to Year 2
Description: All cause HCRU - mean number of outpatient encounters per participant from baseline to year 2 is presented. Physician outpatient office visit is defined by a medical claim with outpatient place of service and an evaluation and management code.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: outpatient encounters
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
outpatient encounters | 18.7 (17.7) | 16.5 (13.2)

34. Secondary Outcome: All Cause HCRU: Mean Number of Medication Visits Per Participant From Baseline to Year 2
Description: All cause HCRU - mean number of medication visits per participant from baseline to year 2 is presented.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: medication visits
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
medication visits | 7.4 (43.1) | 2.9 (5.2)

35. Secondary Outcome: All Cause HCRU: Number of Participants With Inpatient Admission (Yes/No) From Baseline to Year 2
Description: All cause HCRU - number of participants with inpatient admission from baseline to year 2 is presented. Yes: number of participants who experienced inpatient admission; no: number of participants who did not experience inpatient admission.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
Participants
  Yes | 16 | 16
  No | 85 | 86

36. Secondary Outcome: All Cause HCRU: Number of Participants With ER Encounter (Yes/No) From Baseline to Year 2
Description: All cause HCRU - number of participants with ER encounter from baseline to year 2 is presented. Yes: number of participants who experienced ER Encounter; no: number of participants who did not experience ER Encounter.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
Participants
  Yes | 24 | 21
  No | 77 | 81

37. Secondary Outcome: All Cause HCRU: Number of Participants With Outpatient Encounter (Yes/No) From Baseline to Year 2
Description: All cause HCRU - number of participants with outpatient encounter from baseline to year 2 is presented. Physician outpatient office visit is defined by a medical claim with outpatient place of service and an evaluation and management code. Yes: number of participants who experienced outpatient encounter; no: number of participants who did not experience outpatient encounter.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
Participants
  Yes | 97 | 101
  No | 4 | 1

38. Secondary Outcome: Diabetes Related HCRU: Mean Number of Diabetes Related Inpatient Admissions Per Participant From Baseline to Year 2
Description: Diabetes related HCRU - mean number of diabetes related inpatient admissions per participant from baseline to year 2 is presented.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: FAS included all randomized participants analyzed according to the treatment group to which they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for this outcome measure. Analysis is based only on participants with available data for diabetes related HCRU at dedicated study visit including measurements irrespective of whether participants discontinued study drug or not.
Measure: Mean (Standard Deviation); unit: inpatient admissions
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
inpatient admissions | 0.13 (0.37) | 0.19 (0.70)

39. Secondary Outcome: Diabetes Related HCRU: Mean Cumulative Length of Stay for Diabetes Related Inpatient Admissions Per Participant From Baseline to Year 2
Description: Diabetes related HCRU - mean cumulative length of stay for diabetes related inpatient admissions per participant from baseline to year 2 is presented. Cumulative inpatient length of stay is the sum of the length of stay of all diabetes related inpatient admissions a participant experiences from baseline to year 2.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: FAS: all randomized participants analyzed according to treatment group they were assigned at randomization. Overall Number of Participants Analyzed = participants with available data for the outcome measure. Analysis is based only on participants with available data for diabetes related HCRU at dedicated study visit including measurements irrespective of whether participants discontinued study drug/not. It is only calculated for participants with at least 1 diabetes related inpatient admission.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 12 | 12
Days | 4.7 (2.9) | 8.9 (12.1)

40. Secondary Outcome: Diabetes Related HCRU: Mean Number of Diabetes Related ER Encounters Per Participant From Baseline to Year 2
Description: Diabetes related HCRU - mean number of diabetes related ER encounters per participant from baseline to year 2 is presented.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: ER encounters
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
ER encounters | 0.50 (1.49) | 0.17 (0.47)

41. Secondary Outcome: Diabetes Related HCRU: Mean Number of Diabetes Related Outpatient Encounters Per Participant From Baseline to Year 2
Description: Diabetes related HCRU - mean number of diabetes related outpatient encounters per participant from baseline to year 2 is presented. Physician outpatient office visit is defined by a medical claim with outpatient place of service and an evaluation and management code.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: outpatient encounters
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
outpatient encounters | 9.8 (12.9) | 8.1 (5.8)

42. Secondary Outcome: Diabetes Related HCRU: Mean Number of Diabetes Related Medication Visits Per Participant From Baseline to Year 2
Description: Diabetes related HCRU - mean number of diabetes related medication visits per participant from baseline to year 2 is presented.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: medication visits
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
medication visits | 1.4 (2.8) | 1.1 (1.9)

43. Secondary Outcome: Diabetes Related HCRU: Number of Participants With Diabetes Related Inpatient Admission (Yes/No) From Baseline to Year 2
Description: Diabeted related HCRU - number of participants with diabetes related inpatient admission from baseline to year 2 is presented. Yes: number of participants who experienced diabetes related inpatient admission; no: number of participants who did not experience diabetes related inpatient admission.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
Participants
  Yes | 12 | 12
  No | 89 | 90

44. Secondary Outcome: Diabetes Related HCRU: Number of Participants With Diabetes Related ER Encounter (Yes/No) From Baseline to Year 2
Description: Diabeted related HCRU - number of participants with diabeted related ER encounter from baseline to year 2 is presented. Yes: number of participants who experienced diabeted related ER encounter; no: number of participants who did not experience diabeted related ER encounter.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
Participants
  Yes | 18 | 13
  No | 83 | 89

45. Secondary Outcome: Diabetes Related HCRU: Number of Participants With Diabetes Related Outpatient Encounter (Yes/No) From Baseline to Year 2
Description: Diabeted related HCRU - number of participants with diabeted related outpatient encounter from baseline to year 2 is presented. Physician outpatient office visit is defined by a medical claim with outpatient place of service and an evaluation and management code. Yes: number of participants who experienced diabeted related outpatient encounter; no: number of participants who did not experience diabeted related outpatient encounter.
Time Frame: From baseline (less than or equal to 4 weeks prior to the randomization at week 0) to year 2
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 101 | 102
Participants
  Yes | 95 | 97
  No | 6 | 5

46. Secondary Outcome: Number of Participants Who Attained Individualized HbA1c Target at Year 2 (Yes/No)
Description: Number of participants who attained individualized HbA1c target at year 2 is presented. Study physicians set and documented an individualized HbA1c target for participants prior to randomization based on their clinical judgement and knowledge of the participant. Yes: number of participants who achieved individualized HbA1c target attained at year 2; No: number of participants who did not achieve individualized HbA1c target attained at year 2
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 374 | 374
Participants
  Yes | 182 | 129
  No | 192 | 245

47. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) or At Least 1% Point Improvement in HbA1c Compared to Baseline at Year 2 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) or at least 1% point improvement in HbA1c compared to baseline at year 2 is presented. Yes: number of participants who achieved HbA1c less than 7.0% or at least 1% point improvement in HbA1c compared to baseline at year 2; No: number of participants who did not achieve HbA1c less than 7.0% or at least 1% point improvement in HbA1c compared to baseline at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 374 | 373
Participants
  Yes | 274 | 228
  No | 100 | 145

48. Secondary Outcome: Number of Participants With HbA1c Less Than 8.0% (64 mmol/Mol) at Year 1 (Yes/No)
Description: Number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 1 is presented. Yes: number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 1; No: number of participants who did not achieve HbA1c less than 8.0% (64 mmol/mol) at year 1.
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 430 | 462
Participants
  Yes | 344 | 344
  No | 86 | 118

49. Secondary Outcome: Number of Participants With HbA1c Less Than 8.0% (64 mmol/Mol) at Year 2 (Yes/No)
Description: Number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 2 is presented. Yes: number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 2; No: number of participants who did not achieve HbA1c less than 8.0% (64 mmol/mol) at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 374 | 374
Participants
  Yes | 293 | 271
  No | 81 | 103

50. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) and No Further Antidiabetic Medication Intensification After Randomization at Year 1 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) and no further antidiabetic medication intensification after randomization at year 1 is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) and no further antidiabetic medication intensification after randomization at year 1; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) and no further antidiabetic medication intensification after randomization at year 1.
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 430 | 462
Participants
  Yes | 229 | 206
  No | 201 | 254
  Data missing | 0 | 2

51. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) and No Further Antidiabetic Medication Intensification After Randomization at Year 2 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) and no further antidiabetic medication intensification after randomization at year 2 is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) and no further antidiabetic medication intensification after randomization at year 2; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) and no further antidiabetic medication intensification after randomization at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 374 | 373
Participants
  Yes | 186 | 135
  No | 188 | 238

52. Secondary Outcome: Number of Participants With HbA1c Target Attainment Per Healthcare Effectiveness Data and Information Set (HEDIS) Criteria at Year 2 (Yes/No)
Description: Number of participants who achieved HbA1c target attainment per HEDIS criteria (less than 8.0% if age ≥ 65 years or with defined comorbidities, otherwise less than 7.0%) at year 2 is presented. Yes: Number of participants who achieved HbA1c target attainment per HEDIS criteria at year 2; No: Number of participants who did not achieve HbA1c target attainment per HEDIS criteria at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 63 | 52
Participants
  Yes | 43 | 29
  No | 20 | 23

53. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) at Year 1 in Participants With HbA1c >9.0% at Baseline (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) at year 1 in participants with HbA1c >9.0% at baseline is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) at year 1 in participants with HbA1c >9.0% at baseline; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) at year 1 in participants with HbA1c >9.0% at baseline.
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 131 | 122
Participants
  Yes | 41 | 42
  No | 90 | 80

54. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) at Year 2 in Participants With HbA1c >9.0% at Baseline (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) at year 2 in participants with HbA1c >9.0% at baseline is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) at year 2 in participants with HbA1c >9.0% at baseline; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) at year 2 in participants with HbA1c >9.0% at baseline.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 114 | 98
Participants
  Yes | 41 | 28
  No | 73 | 70

55. Secondary Outcome: Number of Participants With HbA1c Less Than 8.0% (64 mmol/Mol) at Year 1 in Participants With HbA1c >9.0% at Baseline (Yes/No)
Description: Number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 1 in participants with HbA1c >9.0% at baseline is presented. Yes: number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 1 in participants with HbA1c >9.0% at baseline; No: number of participants who did not achieve HbA1c less than 8.0% (64 mmol/mol) at year 1 in participants with HbA1c >9.0% at baseline
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 131 | 122
Participants
  Yes | 77 | 67
  No | 54 | 55

56. Secondary Outcome: Number of Participants With HbA1c Less Than 8.0% (64 mmol/Mol) at Year 2 in Participants With HbA1c >9.0% at Baseline (Yes/No)
Description: Number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 2 in participants with HbA1c >9.0% at baseline is presented. Yes: number of participants who achieved HbA1c less than 8.0% (64 mmol/mol) at year 2 in participants with HbA1c >9.0% at baseline; No: number of participants who did not achieve HbA1c less than 8.0% (64 mmol/mol) at year 2 in participants with HbA1c >9.0% at baseline.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 114 | 98
Participants
  Yes | 70 | 53
  No | 44 | 45

57. Secondary Outcome: Percentage Change in Body Weight From Baseline to Year 2
Description: Percentage change in body weight from baseline to year 2 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 389 | 386
Percentage change in body weight | -4.47 (12.204) | -2.68 (7.988)

58. Secondary Outcome: Change in Body Weight (in Pounds) From Baseline to Year 2
Description: Change in body weight (in pounds) from baseline to year 2 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 389 | 386
lbs | -11.1 (24.65) | -6.8 (18.54)

59. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Year 2
Description: Change in SBP from baseline to year 2 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 388 | 386
mmHg | -3.0 (17.03) | -2.8 (16.91)

60. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline to Year 2
Description: Change in DBP from baseline to year 2 is presented.
Time Frame: Baseline (less than or equal to 4 weeks prior to the randomization at week 0), year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 388 | 386
mmHg | -1.9 (10.58) | -1.4 (9.92)

61. Secondary Outcome: Number of Participants With Reported Hypoglycemia Leading to Inpatient Admission or ER Encounter During Year 1 (Yes/No)
Description: Number of participants who reported hypoglycemia leading to inpatient admission or ER encounter during year 1 is presented. Yes: number of participants who reported hypoglycemia leading to inpatient admission or ER encounter during year 1; No: number of participants who did not report hypoglycemia leading to inpatient admission or ER encounter during year 1.
Time Frame: Week 0 to year 1
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 644 | 634
Participants
  Yes | 0 | 0
  No | 644 | 634

62. Secondary Outcome: Number of Participants With Reported Hypoglycemia Leading to Inpatient Admission or ER Encounter During Year 2 (Yes/No)
Description: Number of participants who reported hypoglycemia leading to inpatient admission or ER encounter during year 2 is presented. Yes: number of participants who reported hypoglycemia leading to inpatient admission or ER encounter during year 2; No: number of participants who did not report hypoglycemia leading to inpatient admission or ER encounter during year 2.
Time Frame: Week 0 to year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 644 | 634
Participants
  Yes | 1 | 1
  No | 643 | 633

63. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) Without Experiencing Hypoglycemia Leading to Inpatient Admission or ER Encounter and Body Weight Loss of ≥ 5% Versus Baseline at Year 1 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and body weight loss of ≥ 5% versus baseline at year 1 is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and body weight loss of ≥ 5% versus baseline at year 1; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and body weight loss of ≥ 5% versus baseline at year 1
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 410 | 426
Participants
  Yes | 128 | 68
  No | 282 | 358

64. Secondary Outcome: Number of Participants With Absolute HbA1c Reduction of ≥ 0.5% Without Experiencing Hypoglycemia Leading to Inpatient Admission or ER Encounter and a Body Weight Loss of ≥ 5% Versus Baseline at Year 1 (Yes/No)
Description: Number of participants who achieved absolute HbA1c reduction of ≥ 0.5% without experiencing hypoglycemia leading to inpatient admission or ER encounter and a body weight loss of ≥ 5% versus baseline at year 1 is presented. Yes: number of participants who achieved absolute HbA1c reduction of ≥ 0.5% without experiencing hypoglycemia leading to inpatient admission or ER encounter and a body weight loss of ≥ 5% versus baseline at year 1; No: number of participants who did not achieve absolute HbA1c reduction of ≥ 0.5% without experiencing hypoglycemia leading to inpatient admission or ER encounter and a body weight loss of ≥ 5% versus baseline at year 1.
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 410 | 425
Participants
  Yes | 162 | 79
  No | 248 | 346

65. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) Without Experiencing Hypoglycemia Leading to Inpatient Admission or ER Encounter and Body Weight Loss of ≥ 5% Versus Baseline at Year 2 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and body weight loss of ≥ 5% versus baseline at year 2 is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and body weight loss of ≥ 5% versus baseline at year 2; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and body weight loss of ≥ 5% versus baseline at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 349 | 352
Participants
  Yes | 108 | 76
  No | 241 | 276

66. Secondary Outcome: Number of Participants With Absolute HbA1c Reduction of ≥ 0.5% Without Experiencing Hypoglycemia Leading to Inpatient Admission or ER Encounter and a Body Weight Loss of ≥ 5% Versus Baseline at Year 2 (Yes/No)
Description: Number of participants who achieved absolute HbA1c reduction of ≥ 0.5% without experiencing hypoglycemia leading to inpatient admission or ER encounter and a body weight loss of ≥ 5% versus baseline at year 2 is presented. Yes: number of participants who achieved absolute HbA1c reduction of ≥ 0.5% without experiencing hypoglycemia leading to inpatient admission or ER encounter and a body weight loss of ≥ 5% versus baseline at year 2; No: number of participants who did not achieve absolute HbA1c reduction of ≥ 0.5% without experiencing hypoglycemia leading to inpatient admission or ER encounter and a body weight loss of ≥ 5% versus baseline at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 349 | 351
Participants
  Yes | 136 | 89
  No | 213 | 262

67. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) Without Experiencing Hypoglycemia Leading to Inpatient Admission or ER Encounter and No Body Weight Gain Versus Baseline at Year 1 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and no body weight gain versus baseline at year 1 is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and no body weight gain versus baseline at year 1; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and no body weight gain versus baseline at year 1.
Time Frame: At year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 410 | 426
Participants
  Yes | 199 | 159
  No | 211 | 267

68. Secondary Outcome: Number of Participants With HbA1c Less Than 7.0% (53 mmol/Mol) Without Experiencing Hypoglycemia Leading to Inpatient Admission or ER Encounter and No Body Weight Gain Versus Baseline at Year 2 (Yes/No)
Description: Number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and no body weight gain versus baseline at year 2 is presented. Yes: number of participants who achieved HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and no body weight gain versus baseline at year 2; No: number of participants who did not achieve HbA1c less than 7.0% (53 mmol/mol) without experiencing hypoglycemia leading to inpatient admission or ER encounter and no body weight gain versus baseline at year 2.
Time Frame: At year 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 349 | 352
Participants
  Yes | 159 | 118
  No | 190 | 234

69. Secondary Outcome: Percentage of Medication Possession Ratio (MPR) for Study Drug Medication Adherence For The Two Years of The Study
Description: Percentage of MPR for study drug medication adherence for the two years of the study is presented. Medication adherence referred to a participant's conformance to the provider's recommendation with respect to timing, dosage, and frequency of medication taken during the prescribed length of time. The MPR was used to assess adherence. MPR was calculated as follows: MPR (%) = Sum of days supply for all prescription fills*100/Total number of days in time period. MPR was capped at 100%. MPR was calculated from pharmacy claims data and irrespective of adherence to randomized treatment or changes to antidiabetic treatment.
Time Frame: Week 0 to year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of MPR
Arm/Group | Semaglutide | Standard of Care
Number analyzed (Participants) | 100 | 95
Percentage of MPR | 57.9 (40.5) | 55.7 (38.3)

ADVERSE EVENTS:
Time Frame: Up to year 2 (week 104)
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product or medical device, which does not necessarily have to have a causal relationship to the product or device. The safety population includes all randomized patients initiated on study drug.
Arm/Group | Semaglutide | Standard of Care
All-Cause Mortality (participants affected / at risk) | 9/634 | 9/621
Serious Adverse Events (participants affected / at risk) | 38/634 | 39/621
Other Adverse Events (participants affected / at risk) | 0/634 | 0/621
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=634) | Standard of Care (N=621)
Coronavirus infection (Infections and infestations) | 5 (5) | 5 (6)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Disseminated varicella zoster vaccine virus infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastroenteropancreatic neuroendocrine tumour disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute haemorrhagic ulcerative colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Accidental death (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Breast dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Acinar cell carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Apparent death (General disorders) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03596450/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT03596450/SAP_003.pdf